CLINICAL TRIAL: NCT02289222
Title: 1454GCC: Phase I/II Anti-PD-1 (MK-3475) and IMiD (Pomalidomide) Combination Immunotherapy in Relapsed/Refractory Multiple Myeloma
Brief Title: 1454GCC: Anti-PD-1 (MK-3475) and IMiD (Pomalidomide) Combination Immunotherapy in Relapsed/Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Due to the inclusion of an IMid in combination with pembrolizumab, Study Sponsor terminated the study.
Sponsor: Ashraf Badros (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Ashraf Badros, Sponsor-Investigator, University of Maryland, Baltimore
Organization: University of Maryland, Baltimore (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-00061522; GCC1454
Record Dates: First submitted 2014-10-17; First posted 2014-11-13 (Estimated); Results first posted 2018-08-01 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-11

CONDITIONS: Multiple Myeloma
Keywords: Relapsed/Refractory; MK-3475 & Pomalidomide; Immunotherapy
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — pembrolizumab; pomalidomide; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pomalidomide, Dexamethasone & MK-3475 (Experimental): Pomalidomide is given at standard dose of 4 mg daily orally for 21 days and dexamethasone is given at 40 mg orally weekly. MK3475 will be given as an intravenous infusion at 200 mg every 2 weeks (days 1 and 14).
  Interventions: Drug: MK-3475; Drug: Pomalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: MK-3475 — Anti PD-1 (MD 3475) will be given as an intravenous infusion at 200 mg every 2 weeks.
  Other Names: Generic name: Pembrolizumab - Trade name: Keytruda
Drug: Pomalidomide — Pomalidomide is given at standard dose of 4 mg daily orally for 21 days
  Other Names: Pomalyst, CC-4047, Actimid
Drug: Dexamethasone — Dexamethasone is given at 40 mg orally weekly
  Other Names: Decadron

SUMMARY:
This is an open label trial of Anti PD1/MD-3475, Pomalidomide and dexamethasone. The study will use standard (FDA approved) doses for both pomalidomide and dexamethasone. The experimental drug Anti PD-1 (MK 3475) given on days 1 and 14.

DETAILED DESCRIPTION:
This phase I/II study is focused on patients with relapsed or refractory multiple myeloma. MK-3475 will be given as an intravenous infusion at every 2 weeks. Treatment will be administered on an outpatient basis.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of relapsed and/or refractory MM according to International Myeloma Working Group guidelines (2003)
2. Received two lines of prior therapy that includes an IMiD (lenalidomide or thalidomide) and a proteasome inhibitor (bortezomib and/or carfilzomib) (used either separately or in combination). (a). Prior pomalidomide therapy is permitted, provided the patient achieved at least a partial remission and had not progressed for 3 months after stopping therapy.
3. Measureable disease as defined by the protocol (assessed within 28 days prior to registration).
4. Be willing and able to provide written informed consent/assent for the trial.
5. Be over 18 years of age on day of signing informed consent.
6. Have a performance status of 2 on the ECOG Performance Scale.
7. Demonstrate adequate organ function as defined by the protocol.
8. Female subject of childbearing potential should have a negative serum pregnancy within 72 hours prior to receiving the first dose of study drug.
9. Male subjects should agree to use an adequate method of contraception.

Exclusion Criteria:

1. Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of treatment.
2. Has a diagnosis of immunodeficiency (HIV) or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
3. Has had a prior monoclonal antibody within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
4. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent. (Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.)
5. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or situ cervical cancer that has undergone potentially curative therapy.
6. Has known active central nervous system disease and/or carcinomatous meningitis.
7. Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents.
8. Has evidence of interstitial lung disease or active, non-infectious pneumonitis.
9. Has an active infection requiring systemic therapy.
10. Has a history or current evidence of any condition, therapy, or lab abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
11. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
12. Pregnant or breastfeeding, or expecting to conceive or father children during study participation.
13. Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody as per the protocol.
14. has known active Hepatitis B or Hepatitis C.
15. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies)
16. Has received a live vaccine within 30 days prior to the first dose of trial treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-12-30 (Actual); Primary Completion 2017-08-07 (Actual); Study Completion 2017-08-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf Z Badros, M.B.,Ch.B, Principal Investigator — University of Maryland Greenebaum Cancer Center
Locations (1):
- Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Badros A, Hyjek E, Ma N, Lesokhin A, Dogan A, Rapoport AP, Kocoglu M, Lederer E, Philip S, Milliron T, Dell C, Goloubeva O, Singh Z. Pembrolizumab, pomalidomide, and low-dose dexamethasone for relapsed/refractory multiple myeloma. Blood. 2017 Sep 7;130(10):1189-1197. doi: 10.1182/blood-2017-03-775122. Epub 2017 May 1. PMID 28461396

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the University of Maryland Marlene and Stewart Greenebaum Comprehensive Cancer Center between December 2014 and May 2016.
Period: Overall Study
Arm/Group | Pomalidomide, Dexamethasone & MK-3475
Started | 48
Completed | 48
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pomalidomide, Dexamethasone & MK-3475
Number analyzed (Participants) | 48
Age, Continuous [Median (Full Range); unit: years] | 64 [35 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 46
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 18
  White | 26
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With Adverse Events
Description: Establish the safety and tolerability of Pomalidomide and Dexamethasone in combination with MK-3475
Time Frame: 24 month
Measure: Count of Participants; unit: Participants
Arm/Group | Pomalidomide, Dexamethasone & MK-3475
Number analyzed (Participants) | 48
Participants | 48

2. Secondary Outcome: PD-LI Expression On Myeloma Cells
Description: The identification of a biomarker for response by evaluating PD-1/PDL-1 expression in patients' bone marrow aspirate samples will be analyzed in order to help select patients for future anti-PD-1 therapy. The main exploratory biomarker analysis was to examine potential correlation between expression of PD-1 on T cells and PD-L1 on myeloma cells with clinical outcome using the following parameters: response rate focusing on responses ≥ very good partial response (VGPR) and PFS. SAS software (v.9.4; SAS Institute, Inc, Cary, NC) was used for statistical analyses.
Time Frame: Tissue sample collection will take place before starting study therapy with MK-3475 at baseline and again at time of relapse as defined by the International Myeloma Working Group Response Criteria (Average of up to 24months)
Population: Data were analyzed for 29 samples.
Measure: Count of Participants; unit: Participants
Arm/Group | Pomalidomide, Dexamethasone & MK-3475
Number analyzed (Participants) | 29
Participants
  Negative | 10
  Weak Positive | 6
  Positive | 13

3. Secondary Outcome: Time to Progression Free Survival (PFS)
Description: PFS will be measured in all participants. Survival and PFS functions were estimated using the Kaplan-Meier method. The Cox regression model was used to assess the following plausible risk factors for OS and PFS: age, isotype, number of cycles of therapy, and cytogenetic profile.
Time Frame: PFS assessments will take place after starting study therapy with MD-3475 and will continue until the start of a new anti-neoplastic therapy, disease progression, death, or the end of study up to an average of 24 months.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pomalidomide, Dexamethasone & MK-3475
Number analyzed (Participants) | 48
Months | 17.4 [11.7 to 18.8]

ADVERSE EVENTS:
Time Frame: Reported Adverse Events (AEs) include events starting on or after Day 0 and up to 30 days of receiving the last dose of study medication.
Arm/Group | Pomalidomide, Dexamethasone & MK-3475
All-Cause Mortality (participants affected / at risk) | 2/48
Serious Adverse Events (participants affected / at risk) | 27/48
Other Adverse Events (participants affected / at risk) | 48/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pomalidomide, Dexamethasone & MK-3475 (N=48)
acute coronary syndrome (Cardiac disorders) | 1
heart failure (Cardiac disorders) | 1
cardiac arrest (Cardiac disorders) | 1
adrenal insufficiency (Endocrine disorders) | 1
colitis (Gastrointestinal disorders) | 1
lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
fever (General disorders) | 2
fracture (Injury, poisoning and procedural complications) | 1
hip fracture (Injury, poisoning and procedural complications) | 1
other, bacteremia (Infections and infestations) | 1
skin infection (Infections and infestations) | 1
alanine aminotransferase increased (Investigations) | 1
alkaline phosphatase increased (Investigations) | 1
creatinine increased (Investigations) | 1
hyponatremia (Metabolism and nutrition disorders) | 1
other, meniscus tear (Musculoskeletal and connective tissue disorders) | 1
other, breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
intracranial hemorrhage (Nervous system disorders) | 2
syncope (Nervous system disorders) | 1
urinary retention (Renal and urinary disorders) | 1
bronchitis (Respiratory, thoracic and mediastinal disorders) | 1
dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
lung infection (Respiratory, thoracic and mediastinal disorders) | 9
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1
hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pomalidomide, Dexamethasone & MK-3475 (N=48)
anemia (Blood and lymphatic system disorders) | 26
lymphocyte count decreased (Blood and lymphatic system disorders) | 14
neutrophil count decreased (Blood and lymphatic system disorders) | 30
platelet count decreased (Blood and lymphatic system disorders) | 27
white blood cell decreased (Blood and lymphatic system disorders) | 28
atrial fibrillation (Cardiac disorders) | 3
palpitations (Cardiac disorders) | 6
sinus tachycardia (Cardiac disorders) | 5
ear pain (Ear and labyrinth disorders) | 3
hypothyroidism (Endocrine disorders) | 5
blurred vision (Eye disorders) | 11
abdominal pain (Gastrointestinal disorders) | 6
bloating (Gastrointestinal disorders) | 5
constipation (Gastrointestinal disorders) | 19
diarrhea (Gastrointestinal disorders) | 17
gastroesophageal reflux disease (Gastrointestinal disorders) | 3
nausea (Gastrointestinal disorders) | 10
stomach pain (Gastrointestinal disorders) | 3
vomiting (Gastrointestinal disorders) | 6
chest pain- non cardiac (General disorders) | 3
chest pain- unspecified (General disorders) | 5
chills (General disorders) | 5
edema limbs (General disorders) | 19
fatigue (General disorders) | 23
fever (General disorders) | 5
other, common cold (General disorders) | 10
pain (General disorders) | 3
bruising (Injury, poisoning and procedural complications) | 4
fall (Injury, poisoning and procedural complications) | 10
fracture (Injury, poisoning and procedural complications) | 4
spinal fracture (Injury, poisoning and procedural complications) | 3
skin infection (Infections and infestations) | 4
urinary tract infection (Infections and infestations) | 4
activated partial thromboplastin time prolonged (Investigations) | 4
alanine aminotransferase increased (Investigations) | 15
alkaline phosphatase increased (Investigations) | 7
aspartate aminotransferase increased (Investigations) | 15
blood bilirubin increased (Investigations) | 4
creatinine increased (Investigations) | 19
weight gain (Investigations) | 7
weight loss (Investigations) | 4
hypercalcemia (Metabolism and nutrition disorders) | 7
hyperglycemia (Metabolism and nutrition disorders) | 30
hyperkalemia (Metabolism and nutrition disorders) | 11
hypernatremia (Metabolism and nutrition disorders) | 4
hyperuricemia (Metabolism and nutrition disorders) | 8
hypoalbuminemia (Metabolism and nutrition disorders) | 14
hypocalcemia (Metabolism and nutrition disorders) | 16
hypoglycemia (Metabolism and nutrition disorders) | 8
hypokalemia (Metabolism and nutrition disorders) | 11
hypomagenesemia (Metabolism and nutrition disorders) | 15
hyponatremia (Metabolism and nutrition disorders) | 18
hypohosphatemia (Metabolism and nutrition disorders) | 9
arthralgia (Musculoskeletal and connective tissue disorders) | 12
arthritis (Musculoskeletal and connective tissue disorders) | 4
back pain (Musculoskeletal and connective tissue disorders) | 20
bone pain (Musculoskeletal and connective tissue disorders) | 9
chest wall pain (Musculoskeletal and connective tissue disorders) | 4
flank pain (Musculoskeletal and connective tissue disorders) | 3
generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 4
other, muscle cramp (Musculoskeletal and connective tissue disorders) | 14
pain in extremity (Musculoskeletal and connective tissue disorders) | 16
dizziness (Nervous system disorders) | 23
headache (Nervous system disorders) | 19
other, peripheral neuropathy NOS (Nervous system disorders) | 5
tremor (Nervous system disorders) | 9
anxiety (Psychiatric disorders) | 6
confusion (Psychiatric disorders) | 6
insomnia (Psychiatric disorders) | 13
cough (Respiratory, thoracic and mediastinal disorders) | 8
dyspnea (Respiratory, thoracic and mediastinal disorders) | 26
epitaxis (Respiratory, thoracic and mediastinal disorders) | 6
hiccups (Respiratory, thoracic and mediastinal disorders) | 3
lung infection (Respiratory, thoracic and mediastinal disorders) | 3
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 9
pneumonitis (Respiratory, thoracic and mediastinal disorders) | 6
sore throat (Respiratory, thoracic and mediastinal disorders) | 5
upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 19
hyperhidrosis (Skin and subcutaneous tissue disorders) | 8
other, rash unspecified (Skin and subcutaneous tissue disorders) | 10
pruritis (Skin and subcutaneous tissue disorders) | 10
rash maculopapular (Skin and subcutaneous tissue disorders) | 11
hot flashes (Vascular disorders) | 3
hypertension (Vascular disorders) | 9
hypotension (Vascular disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-07): https://cdn.clinicaltrials.gov/large-docs/22/NCT02289222/Prot_SAP_000.pdf